CLINICAL TRIAL: NCT01928446
Title: CSP #590 - Lithium for Suicidal Behavior in Mood Disorders
Brief Title: Lithium for Suicidal Behavior in Mood Disorders
Acronym: Li+
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: terminated early due to non-safety related DMC recommendations
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 590
Record Dates: First submitted 2013-08-15; First posted 2013-08-26 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder; Bipolar Disorder; Suicide; Suicide, Attempted
Keywords: Lithium; Placebo; Double-blind methods; Clinical Trials, Randomized; Veterans
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Suicide; Suicide, Attempted | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lithium (Experimental): Lithium in the form of extended release lithium carbonate. Subjects will be started on 600 mg/day (300mg bid) until steady state at target plasma levels between 0.6 and 0.8 meq/liter is achieved. The lowest dose will be 300 mg/day. Lithium will be prescribed for the duration of follow-up (1 year).
  Interventions: Drug: Lithium
- Placebo (Placebo Comparator): Placebo tablets will be given to the subjects for the duration of follow-up (1 year). Dose adjustments will mimic the intervention arm of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium in the form of extended release lithium carbonate. Subjects will be started on 600 mg/day (300mg bid) until steady state at target plasma levels between 0.6 and 0.8 meq/liter is achieved. The lowest dose will be 300 mg/day. Lithium will be prescribed for the duration of follow-up (1 year).
  Arms: Lithium
Drug: Placebo — Oral placebo tablets will be administered for the duration of follow-up (1 year).
  Arms: Placebo

SUMMARY:
Observational evidence and findings from clinical trials conducted for other reasons suggest that lithium, a drug used for the treatment of bipolar disorder, and, to a lesser extent, depression, may reduce rates of suicides and suicide attempts. However, this hypothesis has not yet been adequately examined in a randomized clinical trial conducted specifically to test lithium's efficacy in preventing suicides. This clinical trial fills this gap.

This study is feasible within the Department of Veterans Affairs (VA) because it is a large, integrated health system with existing programs for identifying patients at risk for suicide and delivering enhanced services. In VA, approximately 12,000 patients with depression or bipolar disorder survive a suicide attempt or related behavior each year, and 15% of them repeat within one year. Experimental treatment in this study will supplement usual care for major depression or bipolar disorder, as well as VA's standard, enhanced management for patients at high risk.

The investigators will recruit 1862 study participants, from approximately 30 VA Hospitals. Participants will be patients with bipolar disorder or depression who have survived a recent episode of suicidal self-directed violence or were hospitalized specifically to prevent suicide. Randomly, half will receive lithium, and half will receive placebo. Neither the patients nor their doctors will know whether a particular person has received lithium or placebo. The treatment will be administered and the patients will be followed for one year, after which patients will go back to usual care. Recruitment will occur over 3 years.

The investigators are primarily interested in whether lithium leads to increases in the time to the first repeated episode of suicidal behavior, including suicide attempts, interrupted attempts, hospitalizations specifically to prevent suicide, and deaths from suicide. In addition, this study will allow us to explore whether lithium decreases the total number of suicidal behaviors, and whether it has comparable effects on impulsive and non-impulsive behaviors. If there is an effect of lithium, the investigators will be interested in whether or not it could be attributed to improved control of the underlying mental health condition, or, alternatively, whether it represents a direct effect of suicide-related behavior.

DETAILED DESCRIPTION:
Objective: To test the hypothesis that lithium augmentation of enhanced usual care will reduce the rate of repeated episodes of suicidal self-directed violence (repeated suicide attempts, interrupted attempts, hospitalizations specifically to prevent suicide, and deaths from suicide) in participants with bipolar disorder or depression who have survived a recent event.

Background: The hypothesis that lithium can prevent suicide in patients with bipolar disorder and depression is based on data from observational studies and randomized clinical trials conducted to evaluate other outcomes. The question about the effectiveness of lithium for suicide prevention is one of major scientific, clinical, and public health significance. There have been no adequately powered clinical trials conducted specifically to evaluate suicide behaviors as an outcome. Two recent randomized clinical trials failed to recruit adequate numbers of subjects to be conclusive.

The VHA, as a large national healthcare system with an established program for identifying new suicide attempts, evaluating patients for underlying mental health and medical conditions, providing needed services, connecting Veterans to state-of-the-art suicide risk management, and monitoring outcomes is uniquely able to conduct a large scale clinical trial of lithium for suicide prevention.

The rationale for the study is based on the following:

* Data from observational studies and double-blind randomized clinical trials suggest that lithium can prevent suicide-related behaviors in patients with bipolar disorder and major depression.
* The high risk of suicide in Veterans receiving health care services from VHA has persisted despite extensive improvements in mental health services and in programs for suicide prevention.
* Each month, there are over 1,100 unique VHA patients with bipolar disorder or depression who attempt suicide and survive.
* Surviving a suicide attempt is the most powerful known risk factor for death from suicide in VA and elsewhere.
* Approximately 15% of VA survivors reattempt or die from suicide within one year.
* Evaluating rates of reattempts in those who have survived attempts is an established and effective method for testing interventions that may prevent suicide.
* Experimental treatment in CSP-590 would supplement usual care for major depression or bipolar disorder.
* Study procedures for the management of suicide risk would meet or exceed VA standards and requirements.
* Study procedures optimize the safety of lithium, including the potential risk of overdoses, and meet or exceed all published practice standards. The trial will utilize multiple strategies to minimize risks including frequent monitoring and assessment, determination of lithium levels during titration and at steady state, and dispensing medications in limited quantities in blister packs.
* The investigator's survey of VA psychiatrists indicates that the question is clinically important and compelling and that a clinical trial that demonstrated the hypothesized effect would transform the clinical management of suicidality.

Design: Randomized, double-blind, placebo-controlled clinical trial of lithium versus placebo augmentation of enhanced usual care.

Patient population: VHA patients with bipolar disorder or depression who have survived a recent episode of suicidal self-directed violence.

Primary outcome: Time to the first repeated episode of suicidal self-directed violence, including suicide attempts, interrupted attempts, hospitalizations specifically to prevent suicide, and deaths from suicide

Duration: Total study duration will be 4.5 years. Recruitment will occur over 3 years. Participants will be followed for one year.

Sample size calculations and number of sites required: The design of the study is based on testing for a 37% reduction in the rate of repeated suicidal self-directed violence, a figure based on an effect size of approximately 43% observed in recent studies and then allowing for attenuation due to non-adherence. Adjusting for potential data loss due to attrition, 90% statistical power to detect a significant 37% reduction in reattempt rates at 5% overall type I error would require 1862 subjects. With recruitment of 20% of eligible subjects over a three year period, this would require approximately 9310 potentially eligible subjects. Based on current suicide surveillance data, this could be achieved with 29 sites.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran of the United States Armed Forces
* Survived an episode of suicidal self-directed violence (including suicide attempts and interrupted attempts) that occurred within six months of admission to the study, or they were admitted within the past six months to a mental health inpatient unit specifically to prevent suicide
* Have a diagnosis of an affective disorder meeting DSM-IV-TR (2000) criteria for Bipolar I Disorder, Bipolar II Disorder, or current or recurrent Major Depressive Disorder
* Are able and willing to identify one or more family members, friends, or other contacts and give permission for both clinical providers and the Research Team to contact them if the patient cannot be reached
* Are able to provide informed consent
* There is concurrence from the patient's mental health provider about inclusion/exclusion criteria and confirmation of the providers' willingness to work with the research team in managing the patient during the course of the study. The provider responsible for the patient's general medical care has been made aware of the participation
* Must be registered at a VA Medical Center

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Cognitive impairment defined as a Brief Orientation Memory and Concentration Test score > 10
* Lack of decision-making capacity to evaluate the risks versus the benefits of participation as determined by Jeste's brief instrument for assessing decisional capacity, or adjudication of incompetence and the appointment of a guardian or conservator
* Six or more previous lifetime suicide attempts as ascertained through SPAN, reports from family, or patient self-report
* Current or recent (within six months) use of lithium
* History of significant adverse effects of lithium as ascertained through the medical record or self-report
* Unstable medical conditions or specific medical comorbidity:

  * Congestive heart failure by Framingham criteria
  * QTc greater than or equal to 450 ms for men and greater than or equal to 460 ms for women
  * Chronic renal failure defined by national Kidney Foundation Disease Outcome Quality Initiative (KDOQI) criteria
* Any possibility of being pregnant or not on appropriate birth control
* Lactation and breastfeeding
* Concurrent medications:

  * All diuretics except amiloride
  * Haloperidol
  * Clozapine
* Active substance abuse:

  * Active alcohol or opiate dependence requiring medically supervised withdrawal and stabilization
  * Active cocaine, methamphetamine, other stimulant, hallucinogen, or cannabis abuse requiring stabilization
* Enrollment in another randomized interventional clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira R Katz, MD PhD, Study Chair — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (28):
- United States (28):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, NV, Reno, Nevada
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be made available after study closure only to research credentialed Veterans Affairs researchers who submit a valid study question to their IRB of record. A Data Use Agreement will be in effect between the researcher and the coordinating center

REFERENCES:
- [Result] Katz IR, Rogers MP, Lew R, Thwin SS, Doros G, Ahearn E, Ostacher MJ, DeLisi LE, Smith EG, Ringer RJ, Ferguson R, Hoffman B, Kaufman JS, Paik JM, Conrad CH, Holmberg EF, Boney TY, Huang GD, Liang MH; Li+ plus Investigators. Lithium Treatment in the Prevention of Repeat Suicide-Related Outcomes in Veterans With Major Depression or Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):24-32. doi: 10.1001/jamapsychiatry.2021.3170. PMID 34787653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Assessed for eligibility (n=21887).
  2. Signed 1st consent (n=722);
     * Excluded: did not meet inclusion criteria (n= 173).
  3. Signed 2nd consent (n=599);
     * Excluded:
       * not randomized (n=78);
       * assigned to treatment arm, but dropped out prior to receiving Study Meds (n=2).
Period: Overall Study
Arm/Group | Lithium | Placebo
Started | 255 | 264
Completed | 144 (39 subjects stopped study drug but continued with followup) | 125 (23 subjects stopped study drug but continued with followup)
Not Completed | 111 | 139

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium | Placebo | Total
Number analyzed (Participants) | 255 | 264 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.4) | 42.4 (12.4) | 42.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 212 | 225 | 437
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 42 | 77
  Not Hispanic or Latino | 220 | 217 | 437
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 39 | 44 | 83
  White | 185 | 192 | 377
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Time to Event Hazard Rate. Event is a First Repeated Episode of Suicide Related Event, Including Suicide Attempts, Interrupted Attempts and Hospitalizations for Prevention of Attempts.
Description: The primary hypothesis tested is that lithium augmentation of enhanced usual care is superior to enhanced usual care plus placebo for the prevention of repeated episodes of suicidal self-directed violence over time. The investigators posit a one-year repeat rate of 15% in the placebo group and a 37% reduction of events in the intervention group.
  Suicidal self-directed violence includes non-fatal suicide attempts, interrupted attempts (attempts interrupted by patient or by others), hospitalization to prevent suicide and deaths from suicide.
Time Frame: 1 year
Measure: Number; unit: Monthly Hazard rate
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 255 | 264
Monthly Hazard rate | 0.0382 | 0.0348
Statistical Analysis 1: Comparison: Lithium vs Placebo; Model1 - Treatment only: unadjusted for other covariates; Test type: Superiority; p = 0.61, Log Rank; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.77 to 1.55]
Statistical Analysis 2: Comparison: Lithium vs Placebo; Model2 - Treatment only: unadjusted with Site as random Effect; Test type: Superiority; p = 0.67, Log Rank; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.76 to 1.53]

2. Primary Outcome: Number of Compliant Participants With Episode of Self-directed Violence (Per Protocol Analyses)
Description: Compliance is defined as taking 80% or more of study medication over the entire clinical trial.
  Episode of self-directed violence is defined as: First Repeated Episode of Suicide Related Event, Including Suicide Attempts, Interrupted Attempts, Hospitalization to Prevent Suicide and death.
Time Frame: 1 year
Population: Analysis performed for a subset of participants:
  88 of 519 subjects took 80% or more of their study medication (46 on lithium, 42 on placebo) and were considered substantially compliant. Twenty of these subjects had primary outcomes (8 on placebo, 12 on lithium).
Measure: Count of Participants; unit: Participants
Groups:
- Lithium (Compliance Per Protocol); Placebo (Compliance Per Protocol): compliance with study medication, defined as taking 80% or more of their study medication
Arm/Group | Lithium (Compliance Per Protocol) | Placebo (Compliance Per Protocol)
Number analyzed (Participants) | 46 | 42
Participants | 12 | 8
Statistical Analysis 1: Comparison: Lithium (Compliance Per Protocol) vs Placebo (Compliance Per Protocol); Test type: Superiority; p = 0.37, Log Rank; Cox Proportional Hazard = 1.49, 95% CI 2-sided [0.61 to 3.64]

3. Secondary Outcome: Number of Participants With Subtypes of Suicidal Self-directed Violence for All Recurring Events
Description: Subtypes of suicidal self-directed violence:
  1. Self-directed violence;
  2. Interrupted self-directed violence;
  3. Hospitalization to prevent suicide;
  4. Death from suicide - there were too few deaths in the study, making data insufficient to perform analysis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 255 | 264
Participants
  Suicidal self-directed violence | 11 | 10
  Interrupted suicidal self-directed violence | 17 | 11
  Hospitalization to prevent suicide | 34 | 39
  Death from suicide | 1 | 0
  Other | 2 | 2
Statistical Analysis 1: Comparison: Lithium vs Placebo; Model 5: Non-fatal self-directed violence subgroup; Test type: Superiority; p = 0.77, Log Rank; Cox Proportional Hazard = 1.14, 95% CI 2-sided [0.48 to 2.69]
Statistical Analysis 2: Comparison: Lithium vs Placebo; Model 6: Interrupted self-directed violence subgroup; Test type: Superiority; p = 0.22, Log Rank; Cox Proportional Hazard = 1.61, 95% CI 2-sided [0.75 to 3.43]
Statistical Analysis 3: Comparison: Lithium vs Placebo; Model 7: Hospitalization to prevent suicide; Test type: Superiority; p = 0.71, Log Rank; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.58 to 1.45]

ADVERSE EVENTS:
Time Frame: Data collected over 395 days from randomization
Arm/Group | Lithium | Placebo
All-Cause Mortality (participants affected / at risk) | 1/255 | 3/264
Serious Adverse Events (participants affected / at risk) | 99/255 | 90/264
Other Adverse Events (participants affected / at risk) | 193/255 | 166/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=255) | Placebo (N=264)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Serositis (General disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rectal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Antipsychotic drug level increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate abnormal (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (3) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 3 (4)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 2 (3) | 0 (0)
Affective disorder (Psychiatric disorders) | 3 (4) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 2 (6)
Alcoholism (Psychiatric disorders) | 10 (14) | 10 (22)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 2 (3)
Bipolar II disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 7 (8) | 7 (12)
Drug use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 2 (3) | 3 (3)
Major depression (Psychiatric disorders) | 12 (12) | 13 (15)
Mania (Psychiatric disorders) | 1 (1) | 1 (1)
Narcissistic personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 7 (8) | 11 (12)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Substance use disorder (Psychiatric disorders) | 5 (5) | 5 (5)
Substance-induced mood disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 9 (11) | 18 (24)
Suicide attempt (Psychiatric disorders) | 16 (20) | 10 (10)
Suicide threat (Psychiatric disorders) | 0 (0) | 1 (1)
Violence-related symptom (Psychiatric disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bereavement (Social circumstances) | 0 (0) | 1 (2)
Alcohol detoxification (Surgical and medical procedures) | 3 (3) | 4 (7)
Alcohol rehabilitation (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia hiatus repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Mass excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Penile prosthesis insertion (Surgical and medical procedures) | 2 (2) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Wrist surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=255) | Placebo (N=264)
Diarrhoea (Gastrointestinal disorders) | 58 (70) | 41 (50)
Dry mouth (Gastrointestinal disorders) | 12 (12) | 14 (14)
Nausea (Gastrointestinal disorders) | 40 (48) | 26 (30)
Vomiting (Gastrointestinal disorders) | 14 (15) | 6 (7)
Fatigue (General disorders) | 23 (24) | 7 (7)
Thirst (General disorders) | 28 (33) | 23 (24)
Electrocardiogram QT prolonged (Investigations) | 14 (16) | 5 (7)
Glomerular filtration rate decreased (Investigations) | 34 (41) | 22 (32)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 15 (15)
Weight fluctuation (Metabolism and nutrition disorders) | 9 (10) | 21 (22)
Dizziness (Nervous system disorders) | 23 (26) | 14 (16)
Headache (Nervous system disorders) | 30 (32) | 33 (35)
Somnolence (Nervous system disorders) | 18 (18) | 30 (35)
Tremor (Nervous system disorders) | 61 (72) | 19 (19)
Pollakiuria (Renal and urinary disorders) | 22 (25) | 21 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT01928446/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT01928446/SAP_001.pdf
  • Informed Consent Form: Screening ICF (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT01928446/ICF_002.pdf
  • Informed Consent Form: Randomization ICF (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT01928446/ICF_003.pdf